CLINICAL TRIAL: NCT04284501
Title: The Relationship Between Pain Catastrophizing Level, Extreme Sensory Processing Patterns and Headache Severity Among Adolescents With Migraine
Brief Title: Comparing Sensory Modulation, Anxiety and Quality of Life Between Children With Primary Headaches and Healthy Peers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Jacob.genizi, Director Pediatric Neurology Unit, Bnai Zion Medical Center
Other Study IDs: 21-14-BNZ
Record Dates: First submitted 2020-02-16; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: children with Migraine headache
  Interventions: Behavioral: Non
- Control: Healthy children
  Interventions: Behavioral: Non

INTERVENTIONS:
Behavioral: Non — questionnaire

SUMMARY:
Study hypotheses:

1. Children with headaches will show significantly higher sensory reactivity, higher anxiety level and lower quality of life that health controls.
2. Among children with headaches, sensory reactivity will significantly correlate with higher anxiety level and lower quality of life.
3. Among children with headaches quality of life will be predicted by sensory reactivity and anxiety level.

Study significance:

This is one of the first studies to explore the role of sensory reactivity and its relation to the psychological (anxiety) aspects among children and youth with headaches.

Moreover, by using an elaborated point of view this study also measures the interaction between these factors and the child's quality of life.

Referring to this interaction is critical for the intervention process in the meaning of:

(a) helping determine whether pediatric headaches is best conceptualized as a CNS disorder, an emotional disorder, or some hybrid (b) increasing physicians' recognition of headaches pathogenesis and related outcomes, encouraging physicians to refer in the intake and intervention to both children and parents and when needed - to consider mental health services for child/parents. (c) to illuminate the physiological/psychological factors that have the most significant impact on QOL of children with headaches.

Methods:

Participants:

The sample will include 60 children aged 8-18 years. The study group will include 30 children diagnosed with Primary headache - Migraine or TTH. They will be recruited from the pediatric neurological clinic in Bnai-Zion Health Center.

The control group will include 30 children from the community with typical development and no history of chronic headaches or another chronic disease, no ADHD or learning disabilities, matched by age, gender and socio-economic status to the study group.

Inclusion criteria for the study group:

Children with Primary headaches diagnosed as Migraine or TTH between 8-18 years of age.

Exclusion criteria for the sample group Evidence of an inflammatory, anatomic, metabolic, or neoplastic process that explains the subject's symptoms.

DETAILED DESCRIPTION:
Introduction:

Headache is one of the leading chronic conditions bothering children (Newacheck PW 1992) and the most common pain complaint when seeking medical advice (Genizi J 2013), with an evidence for increased incidence of primary headaches in children and adolescents in the last 50 years (Abu-Arefeh I 1994, Goodman JE 1991). As reported by studies, a clear and reliable estimate of the magnitude of the problem has showed that around 60% of the children and adolescents are prone to headache, with attacks of variable frequency (Abu-Arafeh I 2010). The headache begins to emerge during the early years of life, but the disorder usually becomes more evident and frequent from the impact of school life, with a peak around 7 years old (Sillanpa AM 1996).

Migraine and Tension-type headaches (TTH) are the most frequent types of primary headaches in children: The prevalence of migraine is about 10% for girls and about 5% for boys (7% overall), the prevalence of TTH is 0.9% to 24% (Zwart JA 2004, Asuni C 2010).

The diagnosis of primary headaches is mainly supported by anamnestic data and neurological examination (Hershey AD 2010). While Migraine attack has fairly clear diagnostic criteria, with some references to the unique features in children and adolescents, TTH's diagnosis is based almost completely on exclusion criteria, meaning absence of any feature which can fit another type of headache, and no attribution to any special features in children (The International Classification of Headache Disorders: 2nd edition.( ICHD-II)).

Headaches and sensory modulation We didn't find any previous studies on the sensory modulation of patients with headaches, however, children who suffer from primary headaches have an increased risk for emotional and even psychiatric comorbidity such as anxiety and mood disorders (Francesco Margari 2013). In addition, they also have a greater risk of developing psychological disorders in adulthood (Egger HL 1999). Moreover, adolescents who suffer from chronic headaches were found to have more somatic complaints such as abdominal pain and disordered sleep (Genizi J 2013), which can also explains why headaches correlates with a significant reduction in quality of life (Andreas Straube 2013).Aromaa et al. (Aromaa, et al 2000) investigated the pain experiences of headaches in children and their family members and found that Headache children seemed to be more cautious in play and hobbies, because they were afraid of getting hurt. When migraine children were compared with tension- type headache children the following differences were found: headache pain was significantly more intensive among migraine children. They also reported that the mothers of tension-type headache children were more often extremely sensitive to pain compared to mothers of migraine children.

Aromaa et al. found that increased general pain sensitivity proved to characterize children with headache and their parents (Aromaa et al 2000).

Neurophysiological studies have disclosed various abnormalities of spinal, brainstem and cortical responsivity to external innocuous or noxious stimuli in primary headaches: Abnormalities of the habituation/sensitization mechanisms were discovered in migraine. In tension-type headache several researches found some evidence of deficient habituation, and by contrast, other disclosed evidence for sensitization in chronic TTH. Future studies will have to determine whether there is an interaction between abnormal sensory processing and other metabolic abnormalities (Gianluca Coppola 2013).

The interaction between sensory sensitivity and behavioral/ emotional responses:

Sensory hypersensitivity may result from inability to effectively modulate sensory information and to organize this sensory input in order to execute adaptive responses to situational demands (Humphry, 2002). Individuals who are more sensitive to sensory information than others (Aron et al., 1997) often perceive sensory events as noxious and stressful (Bundy et al., 2002). They are more likely to experience depression, anxiety disorders such as social phobia (Neal et al., 2002) and avoidant personality disorder (Johnson et al., 2003, Meyer et al., 2000). They also show high levels of arousal (Pfeiffer et al., 2005).

Dunn's model for sensory processing may provide a possible explanation for the relationship between sensory sensitivity and the behavioral output. Dunn's model outlines the relationship between the person's neurological thresholds and the behavioral response/self regulation continua (Brown et al., 2001, Dunn, 1997). Individuals found in the edges of the interaction of these two continua, exhibit atypical sensory processing patterns.

The neurological threshold refers to the point at which there is enough input to cause a nerve cell or a system to activate (Kandel et al., 2000). The two poles of the neurological threshold continuum are low and high. The low pole indicates that the individual requires low intensity stimuli for neurons to fire and for the individuals to react. The high pole represents individuals who require high intensity stimuli or take longer to react to the same stimuli. The two poles of the self regulation continuum are anchored by passive versus active coping strategies in relation to their thresholds. Individuals who utilize passive strategies, would not counter act to unpleasant stimuli while those individuals who use active strategies act to control the amount and type of sensory input (Dunn, 2007). According to Dunn's model the interaction of these two continua results in four sensory processing patterns. Individuals with high neurological thresholds experience either Low registration (which reflects passive responses) or Sensation Seeking (which reflects an active response). With low registration, people fail to detect or have slow responses to sensation. With sensation seeking, people experience pleasure from rich sensory environment and behaviors that create sensation.

The other two patterns refer to those with low neurological thresholds: Sensation avoiding which is an active strategy in response to a low neurological threshold, and Sensory Sensitivity which reflects a passive pattern in response to low thresholds. People with avoiding patterns engage in behaviors that limit exposure to stimuli, while people with sensory sensitivity experience distractibility and discomfort with sensation (Dunn, 1997).

Referring to the interaction between headaches in research and praxis is of most importance since childhood anxiety disorders often predate depressive disorders and other forms of psychopathology in adolescence and adulthood (Bittner et al., 2007) and are associated with a range of negative consequences in terms of social, academic and personal adjustment (Messer et al., 1994, Waters et al., 2013). Indeed, higher levels of somatic complaints in anxious children are strongly associated with poorer school attendance, school refusal, and poorer academic performance (Hughes et al., 2008). The distress and interference caused by headaches may enhance threat-based cognitions and avoidance behaviour, thus contributing to a vicious cycle of escalating symptom severity and negative functional outcomes (Waters et al., 2013), that may significantly reduce child's quality of life.

The relationship between headaches and quality of life:

Physical complaints as well as mental problems can adversely affect a patient's quality of life (QOL) (Guthrie et al., 2002, Bernklevet al., 2004). Indeed, people with headaches have impaired health-related QOL (Cavallini A1 1995). The relatively high percentage of children with headaches and the associated negative emotional and functional outcomes, emphasize the need to further explore additional involved factors that may contribute to the headaches outcomes.

One of the factors that may be found among patients with headaches is sensory hypersensitivity, which is part of a wider concept called sensory processing disorders that include extreme hyper or hypo sensitivity to sensations. However, the knowledge about sensory processing patterns of children and youth with headaches as well as its interaction with child's emotional aspects and quality of life is scarce.

Elaborating this knowledge may assist in focusing intervention on child and family specific organic and emotional needs and thus optimize intervention outcomes and elevate quality of life.

Study hypotheses:

1. Children with headaches will show significantly higher sensory reactivity, higher anxiety level and lower quality of life that health controls.
2. Among children with headaches, sensory reactivity will significantly correlate with higher anxiety level and lower quality of life.
3. Among children with headaches quality of life will be predicted by sensory reactivity and anxiety level.

Study significance:

This is one of the first studies to explore the role of sensory reactivity and its relation to the psychological (anxiety) aspects among children and youth with headaches.

Moreover, by using an elaborated point of view this study also measures the interaction between these factors and the child's quality of life.

Referring to this interaction is critical for the intervention process in the meaning of:

(a) helping determine whether pediatric headaches is best conceptualized as a CNS disorder, an emotional disorder, or some hybrid (b) increasing physicians' recognition of headaches pathogenesis and related outcomes, encouraging physicians to refer in the intake and intervention to both children and parents and when needed - to consider mental health services for child/parents. (c) to illuminate the physiological/psychological factors that have the most significant impact on QOL of children with headaches.

Methods:

Participants:

The sample will include 200 children aged 5- 18 years. The study group will include 100 children diagnosed with Primary headache - Migraine or TTH. They will be recruited from the pediatric neurological clinic in Bnai-Zion Health Center.

The control group will include 100 children from the community with typical development and no history of chronic headaches or another chronic disease, no ADHD or learning disabilities, matched by age, gender and socio-economic status to the study group.

Inclusion criteria for the study group:

Children with Primary headaches diagnosed as Migraine or TTH between 4-18 years of age.

Exclusion criteria for the sample group Evidence of an inflammatory, anatomic, metabolic, or neoplastic process that explains the subject's symptoms.

Assessments:

Questionnaires completed by the parents:

Health and demographic questionnaire - that will include socio-demographic information about the child and his/her family as well as information about child's development and health status. This questionnaire will be filled by the parents and will serve for assuring inclusion criteria.

Short Sensory Profile (SSP) (McIntosh DN, 1999): This is a shorter version of the Sensory Profile (Dunn W, 1999), an instrument used for evaluating sensory processing abilities. The shorter caregiver report measure is comprised of the 38 items that demonstrated the highest discriminative power of atypical sensory processing among all the items from the longer version of the Sensory Profile. The seven sections of the SSP found in a normative sample are Tactile Sensitivity; Test/Smell Sensitivity; Movement Sensitivity; Under-responsive/Seeks Sensation; Auditory Filtering; Low Energy/Weak; and Visual/Auditory Sensitivity. Internal consistency of the sections within the scale ranged from .70 to .90 (Dunn W, 1999). Internal validity correlations for the sections ranged from .25 to .76 and were all significant at p<.01. Initial studies of the validity of the SSP demonstrated discriminate validity of >95% in identifying children with and without sensory modulation difficulties (McIntosh DN, 1999). Items are scored on a five-point scale. Both section scores and a total score are recorded on the SSP. The possible range of raw scores on the total scale is 38 to 190, with higher scores (155-190) reflecting normal performance. A score of 142-154 reflects a probable difference in performance, while a score of 38-141 reflects a definite difference in performance (Dunn W, 1999). Time to complete the questionnaire: 10 minutes.

Questionnaires completed by the children:

State-Trait Anxiety Inventory (STAI) for children - It is comprised of separate, self-report scales for measuring two distinct anxiety concepts: state anxiety (S-Anxiety) and trait anxiety (T-Anxiety). The STAIC is similar in conception and structure to the which provides measures of anxiety for adolescents and adults (Spielberger CD et al., 1970). While especially constructed to measure anxiety in nine- to twelve-year old children, the STAIC may also be used with younger children with average or above reading ability and with older children who are below average in ability.

Pediatric Quality of Life Inventory (Varni JW et al., 2006)- This is a short version of the World Health Quality of Life questionnaire. It includes 23 statements which evaluate the person's perception about his/her quality of life in regard to: physical health; psychological health; social relationship and environment. Each statement is rated on a 0-4 scale which reflects the person's satisfaction from the content appearing in each statement (0=never; 4 = always). Internal consistency of the questionnaire ranted between 0.7-0.9. The questionnaire was found to differentiate between children with chronic health conditions and healthy controls (t=-7.29; p=.001) (Varni JW et al., 2001).

Ped MIDAS The Migraine Disability Assessment (MIDAS) questionnaire was developed to measure the effect migraine headaches have on your daily function. It tries to determine how many days of the child's life were affected to the point that he was unable to function in a way to which he was accustomed. MIDAS takes into account the past three months when asking the questions. It was later adapted for children and given the label "PedMIDAS" (as in, pediatric). (Hershey AD, 2001) The PedMIDAS questionnaire also includes two other pieces of information that are not used for calculating the child's disability score, but that give one more way to illustrate to his or her health care provider how migraines affect your child's life. It asks simply for an assessment of the headache frequency and severity for him or her. The child's health care provider will take this information and couple it with the score to try and gain a more accurate picture of how migraines are affecting your child (Hershey AD, 2004).

Procedure:

After receiving the ethical approvals for conducting this study by the Helsinki committee and by the ethical board of the Faculty of Social Welfare and Health Sciences at the University of Haifa, advertisements published in the clinics will call parents and children to participate in a study about the relationship between child's headaches, sensory sensitivity, anxiety and quality of life.

Participants from the study group, who will answer the inclusion criteria will be invited to the clinic. While the physician will diagnose the child, the parents will fill the questionnaires. Following the physician examination, each child will be asked to complete the STAI and the Peds-QL in a quite room with the research assistant.

For the control group we will use information from previous studies.

Data Analysis:

Descriptive statistics will profile the socio-demographic and the scores of all dependent variable, in each group. Significance of differences between groups will be examined by MANOVA. Correlations between the dependent parameters will be examined by Pearson correlation test. The ability of the dependent parameters to predict QOL will be examined by Linear Regression Test.

The level of significance will be set on p≤.005.

ELIGIBILITY:
Inclusion criteria for the study group:

Children with Primary headaches diagnosed as Migraine or TTH between 8-18 years of age.

Exclusion criteria for the sample group Evidence of an inflammatory, anatomic, metabolic, or neoplastic process that explains the subject's symptoms.

Ages: 8 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-08-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Extreme sensory processing patterns in the Short Sensory Profile questionnaire | 10years
  The Short Sensory Profile (SSP)(26)- This parent report evaluated children's sensory processing patterns, as expressed in all sensory modality and in daily living situations (for example: "will only eat certain tastes"; "reacts emotionally or aggressively to touch"). The Parent scores their childs' response to sensory stimuli on a 5 point Likert scale, where 1 represents "always" and 5 "never". Seven subtests are scored: tactile sensitivity, taste/smell sensitivity, sensitivity to movement, visual/auditory sensitivity and auditory filtering, as well as a total score which ranges between 38 to 190. Higher scores (155-190) reflect typical/normal performance. A score between 142-154 reflects a probable difference in performance while a score between 38-141 reflects a definite difference in performance

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Genizi, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bani Zion, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided